CLINICAL TRIAL: NCT01951235
Title: A Dose-ranging, Randomized, Double-blind, Placebo-controlled, Parallel-group, Multi-center Study of the Efficacy and Safety of 4 Doses of Imeglimin After 24 Weeks of Treatment in Subjects With Type 2 Diabetes Mellitus.
Brief Title: A Study of the Efficacy and Safety of 4 Doses of Imeglimin After 24 Weeks of Treatment in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Poxel SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PXL008-008; 2012-004045-33 (EudraCT Number)
Record Dates: First submitted 2013-09-19; First posted 2013-09-26 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-07

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — imeglimin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Imeglimin (Dose 1) (Experimental)
  Interventions: Drug: Imeglimin
- Imeglimin (Dose 2) (Experimental)
  Interventions: Drug: Imeglimin
- Imeglimin (Dose 3) (Experimental)
  Interventions: Drug: Imeglimin
- Imeglimin (Dose 4) (Experimental)
  Interventions: Drug: Imeglimin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Imeglimin
  Arms: Imeglimin (Dose 1); Imeglimin (Dose 2); Imeglimin (Dose 3); Imeglimin (Dose 4)
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study will assess the efficacy and safety/tolerability of 4 doses of Imeglimin versus placebo. The study will be performed in subjects with type 2 diabetes either naive of treatment or previously treated with an oral monotherapy excluding thiazolidinedione.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has given written informed consent
2. Male and female type 2 diabetic subjects, either naïve of antidiabetic agents or treated with an oral anti-diabetic monotherapy.
3. Body mass index (BMI) : ≥ 24 to ≤ 40 kg/m²
4. HbA1c criteria: ≥ 7% and ≤ 9.5%
5. Creatinine clearance ≥ 50 mL/[min*1.73 m2] at Screening Visit
6. Effective contraception for women of child bearing potential

Exclusion Criteria:

1. Any disease which in the investigator's opinion would exclude the subject from the study
2. Acute cardiovascular event within 3 months before randomization
3. Uncontrolled high blood pressure
4. Impairment of hepatic function
5. History of drug-induced Torsades de Pointes or a marked baseline prolongation of the QTc interval
6. Pregnancy or lactation
7. Use of any non-permitted medication
8. Positive screen for viral hepatitis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2013-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | Baseline and week 24

SECONDARY OUTCOMES:
Safety will be assessed by the incidence of adverse events (AEs), physical examination, relevant changes on laboratory tests, vital signs, and 12-lead electrocardiograms (ECG) | Baseline to week 24

CONTACTS AND LOCATIONS:
Overall Officials: Valdis Pirags, MD, Principal Investigator — P. Stradins Clinical University Hospital
Locations (1):
- Pauls Stradins Clinical University Hospital, Riga, Latvia